CLINICAL TRIAL: NCT00451334
Title: Safety and Efficacy of Using GlucoSat Technology For Non-Invasive Glucose Measurement
Acronym: GS
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Other Study IDs: GS-01
Record Dates: First submitted 2007-03-22; First posted 2007-03-23 (Estimated); Last update posted 2007-03-23 (Estimated); Status verified 2006-11

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Time Perspective: Other
Oversight: Data Monitoring Committee: No

SUMMARY:
This study is a prospective, open label, controlled, single center study. 40 patients will be recruited for the study, according to patients' inflow and meeting eligibility criteria.

Primary Goal

* To evaluate the safety of the GlucoSat technology as a non-invasive blood glucose level measurement technology.

Secondary Goal

* To assess the efficacy of the GlucoSat technology as a non-invasive blood glucose level measurement technology.

DETAILED DESCRIPTION:
Primary Endpoint Parameter

• Primary study endpoint will be to establish the safety of using the GlucoSat technology as a non-invasive glucose level measurement technology. Safety will be established by paucity of adverse events. Adverse Events occurrence will be documented throughout the study.

Secondary Endpoint Parameters

Efficacy of the GlucoSat technology will be assessed by:

* Proving the accuracy and precision of the GlucoSat technology by comparing the glucose level measured by the GlucoSat device to the glucose level observed by any certified for clinics invasive device. Inter device variability should be within 15%.
* Patient satisfaction questionnaire.
* Physician satisfaction will be assessed by questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Male/Female aged 18 and up.
* Subject was diagnosed as a diabetes patient or healthy subject.
* Subject able to comprehend and give informed consent for participation in this study.
* Signed Informed Consent Form

Exclusion Criteria:

* Pregnancy or breast feeding.
* Patients treated with steroid.
* Concomitant Coumadin use
* Recent (within the last 3 months) myocardial infarction or CVA (stroke).
* Any chronic unstable disease within the last 3 months.
* Acute bleeding disorders.
* HIV positive.
* Hepatitis B/C positive.
* BMI>37
* Needing emergency surgery
* Known cognitive or psychiatric disorder
* Physician objection
* Concurrent participation in any other clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40

CONTACTS AND LOCATIONS:
Overall Officials: Shai Efrati, MD, Principal Investigator
Locations (1):
- Assaf-Harofeh Medical Center, Zrifin, Israel